CLINICAL TRIAL: NCT02335021
Title: The Effect of Artificial Sweeteners (AFS) on Sweetness Sensitivity, Preference and Brain Response in Adults
Acronym: AFS-adult
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 0405026766-2
Record Dates: First submitted 2014-10-24; First posted 2015-01-09 (Estimated); Last update posted 2019-09-26 (Actual); Status verified 2019-09

CONDITIONS: Impairment of Oral Perception; Insulin Resistance
MeSH Terms: conditions — Insulin Resistance | interventions — trichlorosucrose; Sucrose; maltodextrin

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Sucralose (Experimental): Participants will rate sweetness, sourness, saltiness, bitterness and umami intensity of various taste stimuli. Next they will consume a flavored beverage with sucralose.
  Interventions: Dietary Supplement: Sucralose
- Sucrose (Experimental): Participants will rate sweetness, sourness, saltiness, bitterness and umami intensity of various taste stimuli. Next they will consume a flavored beverage with sucrose.
  Interventions: Dietary Supplement: Sucrose
- Sucralose + maltodextrin (Experimental): Participants will rate sweetness, sourness, saltiness, bitterness and umami intensity of various taste stimuli. Next they will consume a flavored beverage with Splenda + maltodextrin .
  Interventions: Dietary Supplement: Sucralose + maltodextrin
- Sucralose + Sucrose (Experimental): Participants will rate sweetness, sourness, saltiness, bitterness and umami intensity of various taste stimuli. Next they will consume a flavored beverage with Splenda + sucrose.
  Interventions: Dietary Supplement: Sucralose + Sucrose

INTERVENTIONS:
Dietary Supplement: Sucralose — 2 packets per 12 fl oz
  Arms: Sucralose
Dietary Supplement: Sucrose — equisweet to sucralose
  Arms: Sucrose
Dietary Supplement: Sucralose + maltodextrin — sucralose plus equicaloric (to sucrose) maltodextrin
  Arms: Sucralose + maltodextrin
Dietary Supplement: Sucralose + Sucrose — half the amount of sucralose plus equicaloric sucrose
  Arms: Sucralose + Sucrose

SUMMARY:
The purpose of this study is to investigate the effects of dietary exposure to artificial sweeteners on taste sensitivity, preference and brain response in adults. The investigators hypothesize that dietary exposure to artificial sweeteners (sucralose) will decrease sensitivity to taste, shift preference of sweet and savory taste to a higher dose, and reduce brain response in amygdala to sweet taste compared to sucrose.

DETAILED DESCRIPTION:
We aim to identify neural factors that contribute to taste intensity perception in humans and to determine environmental mechanisms that contribute to variation in taste sensitivity. Significant controversy surrounds the possibility that consumption of artificial sweeteners (AFS) leads to weight gain. Given that the five FDA approved AFSs are found in thousands of foods (Yang 2010) this marks a clear and significant gap in knowledge. Our preliminary data demonstrate a 3-fold decrease in sweet taste sensitivity following consumption of a beverage sweetened with two packets of Splenda for just 10 days. These data provide strong evidence that repeated exposure to sucralose reduces perception of sweet taste intensity, most likely by down-regulation of the sweet taste receptor. Therefore, it is imperative that we gain a greater understanding of the physiological consequences of AFS, since alterations in sweet taste perception, metabolism and brain reward that occur in response to AFS exposure may promote weight gain.

ELIGIBILITY:
Inclusion Criteria:

* Healthy
* Fluent in English
* Right handed

Exclusion Criteria:

* History of oral nerve damage,
* presence of known taste or smell disorder,
* food allergies or sensitivities (for example nuts, lactose, artificial sweeteners),
* history of CNS disease,
* diabetes,
* history of DSM-IV major psychiatric disorder,
* including alcohol and substance abuse,
* chronic use of medication that may affect taste,
* conditions that may interfere with gustatory or olfactory perception (colds, seasonal allergies,
* recent smoking history),
* aberrant stimulus ratings,
* contra-indication for fMRI,
* uncomfortable swallowing in supine position,
* discomfort or anxiety associated with insertion an intravenous catheter,
* regular artificial sweetener use.

Ages: 23 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 97 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2019-04-24 (Actual); Study Completion 2019-04-24 (Actual)

PRIMARY OUTCOMES:
Ratings of taste sensitivity | up to one week after intervention
  general labeled magnitude scale ratings of taste intensity

SECONDARY OUTCOMES:
Ad libitum food intake | up to one week after intervention
  amount of Mac&Cheese consumed
brain response to taste stimuli | up to one week after intervention
  BOLD response as measured by fMRI

CONTACTS AND LOCATIONS:
Overall Officials: Dana M Small, Principal Investigator — Yale University
Locations (1):
- Yale University, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be publicly shared at publication of manuscript.
Time Frame: De-identified data will be publicly shared at publication of manuscript (anticipated in 2019). Data will be available indefinitely, or at least as long as the hosting platform is available.